CLINICAL TRIAL: NCT04755023
Title: Primary Chemotherapy by BCNU-TMZ Combination in Newly Diagnosed Anaplastic Oligodendrocytic Tumors: Phase II Trial With Translational Molecular Analysis
Acronym: TEMOBIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-30
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Oligodendroglioma; Oligoastrocytoma
Keywords: chemotherapy; BCNU-Temozolomide; radiotherapy
MeSH Terms: conditions — Oligodendroglioma; Astrocytoma | interventions — Carmustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Administration of 6 cycles of chemotherapy
  Interventions: Drug: Bis-Chloroethyl-Nitroso-Urea (BCNU) withTemozolomide

INTERVENTIONS:
Drug: Bis-Chloroethyl-Nitroso-Urea (BCNU) withTemozolomide — Chemotherapy (BCNU) will be delivered at Day 1. between day 1 and day 5, temolozomide will be administered . One cycle is planned every 6 weeks until 6 cycles.

SUMMARY:
The first-line treatment of anaplastic oligodendrogliomas, radiotherapy exclusive or combined with PCV, will be defined by the pending results of phase III of the EORTC.

If the phase II study proposed here achieves its objective, it may help define a new treatment regimen that will be compared to the standard arm from phase III of the EORTC.

In addition, this study, by prospectively testing the predictive value of 1p and 19q deletions and of REGF amplification, may allow characterization of patients using these markers. If validated, this characterization can constitute a key element in any therapeutic evaluation (patient stratification), and potentially a major tool for medical decision support in these tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven oligodendroglioma or anaplastic oligoastrocytoma, newly diagnosed, resulting or not from a low grade glioma
* Tumor with measurable contrast enhancement (at least 15 mm in diameter)
* Surgical procedure limited to a biopsy or partial excision
* In the event of partial excision, an early postoperative check-up (<72 hours) performed at best by MRI, if not by CT, is required.
* Time between surgery and inclusion less than or equal to one and a half months (45 days)
* Age> 18 years old; <70
* Karnofsky index> 60
* Stable or reduced dose of corticosteroids in the 15 days prior to inclusion
* Polynuclear neutrophils> 1500; platelets> 100,000
* Bilirubin <1.25 x UNL; SGOT, SGPT, PAL <2.5 x UNL
* Absence of serious uncontrolled pathology
* Patient having received and understood the information and having signed the consent

Exclusion Criteria:

* Presence of GBM foci within the tumor
* Absence of evaluable residue after surgery
* Previous chemotherapy or radiotherapy
* Unsatisfactory expected monitoring conditions
* Pregnant or breastfeeding woman; lack of effective contraception if of childbearing age
* History of malignant disease (with the exception of CIS of the cervix and basal cell cancer)
* Contraindications related to the examination of the I.R.M.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-12-21 (Actual); Primary Completion 2009-03-15 (Actual); Study Completion 2010-12-15 (Actual)

PRIMARY OUTCOMES:
Objective response rate of the BCNU-TMZ combination administered before radiotherapy | At the end of Cycle 2 (each cycle is 28 days)
  In oligodendrogliomas and anaplasic oligoastrocytomas as the first line of treatment
Objective response rate of the BCNU-TMZ combination administered before radiotherapy | At the end of Cycle 4 (each cycle is 28 days)
  In oligodendrogliomas and anaplasic oligoastrocytomas as the first line of treatment
Objective response rate of the BCNU-TMZ combination administered before radiotherapy | At the end of Cycle 6 (each cycle is 28 days)
  In oligodendrogliomas and anaplasic oligoastrocytomas as the first line of treatment
Objective response rate of the BCNU-TMZ combination administered before radiotherapy | 1 month after radiotherapy
  In oligodendrogliomas and anaplasic oligoastrocytomas as the first line of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique - Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No